CLINICAL TRIAL: NCT04272671
Title: Implementation of a De-prescribing Medication Program to Evaluate Falls in Older Adults
Brief Title: De-prescribing Program to Evaluate Falls in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-2920; CE 18-004 (Other: UNC)
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Opioid-Related Disorders; Benzodiazepine-Related Disorders; Falls Injury
Keywords: De-Prescribing; Falls in Older Adults; Benzodiazepines; Opioid
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: This trial uses a cluster-randomized pragmatic design wherein clinics are randomized into intervention and control, and all patients receiving care from those clinics are categorized into intervention or control based on their clinic's participation.
Masking Description: As this is a pragmatic design, there will be no blinding for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Educational Intervention Arm (Experimental): The intervention arm will receive educational material that enhances the standard of care for deprescribing opioids and BZDs.
  Interventions: Other: Educational Intervention
- Ususal Care (Control Arm) (No Intervention): Control group will receive standard of care

INTERVENTIONS:
Other: Educational Intervention — The intervention has the following components: 1) alerts given to providers to identify patients taking opioids or benzodiazepines (BZD) and therefore at risk for falls; 2) educational materials to inform providers on best practices for de-prescribing opioids and BZDs in patients at risk; and 3) recommendations on de-prescribing provided by a consultant pharmacist. Impact of the intervention will be evaluated using pre-post surveys evaluating changes in providers' knowledge, confidence, and skills as well as information from the EHR to evaluate impact of the intervention on de-prescribing opioids and BZDs.
  Arms: Educational Intervention Arm

SUMMARY:
Purpose: The proposed study will implement and evaluate the effect of an opioid and benzodiazepine (BZD) de-prescribing intervention on falls risk in older adults.

Participants: Outpatient clinics with older adult patients, healthcare providers, older adult patients

Procedures (methods): In this proposed study, there will be 10 primary care clinics randomly assigned to the intervention arm and 10 primary care clinics randomly assigned to the control arm. In the first phase of this study, patient and provider focus groups will be used to inform the development of the intervention which will be tested during the active trial phase. The intervention has the following components: 1) alerts given to providers to identify patients taking opioids or benzodiazepines (BZD) and therefore at risk for falls; 2) educational materials to inform providers on best practices for de-prescribing opioids and BZDs in patients at risk; and 3) recommendations on de-prescribing provided by a consultant pharmacist. Impact of the intervention will be evaluated using pre-post surveys evaluating changes in providers' knowledge, confidence, and skills as well as information from the electronic health record (EHR) to evaluate impact of the intervention on de-prescribing opioids and BZDs.

DETAILED DESCRIPTION:
Falls among older adults is costly and dangerous. Observational studies show consistent associations between falls and certain medications. It is widely accepted that falls-related morbidity and mortality could be reduced if systems were in place to identify falls risks and intervene to reduce the risks identified. In this study, health care professionals (HCPs) within UNC outpatient clinics will be alerted to patients on high-risk medications and provide team-based interventions to maximize the success of falls education and medication deprescribing.

This deprescribing intervention will focus specifically on opioids and benzodiazepines (BZDs) in patients 65 years of age and older since these medications have high susceptibility to negative cognitive effects in older adults and contribute to a higher risk of falls. This study will identify factors affecting the adoption, effective implementation, and maintenance of a deprescribing program focused on opioids and BZDs with the intent of reducing falls.

ELIGIBILITY:
Inclusion Criteria:

* UNC HealthCare clinic providing primary care services
* age at least 65 years old
* taking at least one chronic opioid or one chronic benzodiazepine medication

Exclusion Criteria:

* Clinics that do not provided primary care services
* Patients who exhibit signs of cognitive impairment or speech/hearing deficits that make obtaining informed consent and completing data collection activities difficult
* Patients undergoing active cancer treatment, receiving hospice care, or living in a skilled nursing facility
* Non-English speaking patients will be excluded from participating in the patient focus group.
* Participants who do not wish to be audio-recorded during focus group

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Changes in Opioid and/or BZD use | 1 year pre-intervention, 1 year post intervention
  Changes in opioid use will be measured using milligram morphine equivalents per day and benzodiazepine use will be measure using lorazepam or diazepam equivalents per day

SECONDARY OUTCOMES:
Frequency of Falls | 1 year pre-intervention, 1 year post intervention
  evaluating the educational impact on opioid and BZD deprescribing in relation to falls looking at the rate of falls 1 year per-intervention and the rate at completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Ferreri, Principal Investigator — University of North Carolina, Chapel Hill; Jan Busby-Whitehead, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: Made available for 12-36 months following the publication of the primary manuscript from the trial.
Access Criteria: Contact study primary investigator at stefanie_ferreri@unc.edu

REFERENCES:
- [Derived] Niznik J, Ferreri SP, Armistead L, Urick B, Vest MH, Zhao L, Hughes T, McBride JM, Busby-Whitehead J. A deprescribing medication program to evaluate falls in older adults: methods for a randomized pragmatic clinical trial. Trials. 2022 Apr 4;23(1):256. doi: 10.1186/s13063-022-06164-5. PMID 35379307